CLINICAL TRIAL: NCT07112014
Title: Development of Gastrointestinal Symptoms in Patients With Anorexia Nervosa and Bulimia Nervosa During Weight Rehabilitation Over Time, Depending on the Nutritional Strategy
Acronym: GastroRehab
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: GastroRehab
Record Dates: First submitted 2025-07-15; First posted 2025-08-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: gastrointestinal symptoms; gastrointestinal health; dietary regime; psychological health; vegetarian diet; vegan diet; balanced diet; energy intake
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with anorexia nervosa and bulimia nervosa: The study population includes patients with anorexia nervosa (AN) and bulimia nervosa (BN) who participate in an established, multi-week inpatient treatment program aimed at weight rehabilitation and normalization of eating behavior at the Eating Disorder Center of the Klinik Lüneburger Heide in 29549 Bad Bevensen, Germany. The diagnostic and treatment of the patients is as usual. These data, including detailed data on dietary intake, are used for the study. Additionally, information on gastrointestinal sympoms are assessed upon admission and discharge and weekly during the inpatient stay. The outcomes will be analyzed seperately for patients with anorexia nervosa and bulimia nervosa.

SUMMARY:
This prospective observational study investigates the development of gastrointestinal (GI) symptoms in patients with anorexia nervosa (AN) and bulimia nervosa (BN) during multi-week inpatient weight rehabilitation. The study explores how the predominant nutritional strategy-flexitarian, vegetarian, or vegan-relates to changes in GI symptoms over the course of treatment. In addition to diet, the study examines how weight gain and other clinical, psychological, and demographic factors influence the trajectory of GI symptoms. Patients complete weekly questionnaires assessing GI symptoms as part of routine care at the Eating Disorder Center of the Klinik Lüneburger Heide, Germany. Further data are drawn from standard clinical assessments, including body weight, body composition, and psychometric instruments. The primary outcome is the change in GI symptom severity (measured via the GSRS score) from admission to discharge, analyzed in relation to dietary pattern and weight development. Secondary analyses will explore symptom progression over time, group differences between AN and BN, and predictors of GI symptom improvement, including dietary intake, baseline psychological status, symptom change, weight trajectory, and treatment duration. The outcomes will be analyzed separately for AN and BN. The study aims to recruit approximately 150 patients with AN and 35-40 with BN. Inclusion requires a diagnosis of AN (any subtype) or BN, age over 12 years, clinical stability, and the ability to provide informed consent. The findings aim to inform evidence-based dietary recommendations for individuals with eating disorders who experience significant GI symptoms during nutritional rehabilitation.

DETAILED DESCRIPTION:
This prospective observational study investigates the development of gastrointestinal (GI) symptoms in patients with anorexia nervosa (AN) and bulimia nervosa (BN) during multi-week inpatient weight rehabilitation. The study explores how the predominant nutritional strategy-flexitarian, vegetarian, or vegan-relates to changes in GI symptoms over the course of treatment. In addition to diet, the study examines how weight gain and other clinical, psychological, and demographic factors influence the trajectory of GI symptoms. Patients complete weekly questionnaires assessing GI symptoms as part of routine care at the Eating Disorder Center of the Klinik Lüneburger Heide, Germany. Further data are drawn from standard clinical assessments, including body weight, body composition, and psychometric instruments. The primary outcome is the change in GI symptom severity (measured via the GSRS score) from admission to discharge, analyzed in relation to dietary pattern and weight development. Secondary analyses will explore symptom progression over time, group differences between AN and BN, and predictors of GI symptom improvement, including dietary intake, baseline psychological status, symptom change, weight trajectory, and treatment duration. The study aims to recruit approximately 150 patients with AN and 35-40 with BN. Inclusion requires a diagnosis of AN (any subtype) or BN, age over 12 years, clinical stability, and the ability to provide informed consent. The findings aim to inform evidence-based dietary recommendations for individuals with eating disorders who experience significant GI symptoms during nutritional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with anorexia nervosa (all subtypes)
* patients diagnosed bulimia nervosa

Exclusion Criteria:

* patients that are medically unable to fill out a short questionnaire on a weekly base.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Anorexia nervosa and Bulimia nervosa. All subtypes will be included.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptoms | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  Score of the Gastrointestinal Symptom Rating Scale assessed upon admission and discharge (two time points), in relation to the predominant dietary pattern (>80% during the rehabilitation phase), defined as flexitarian, vegetarian, or vegan and body weight development. The Gastrointestinal Symptom Rating Scale is a validated questionnaire : Svedlund J, Sjödin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. (1988) 33(2):129-34. doi: 10.1007/BF01535722. The primary outcome is analyzed seperately for patients with anorexia nervosa and bulimia nervosa.

SECONDARY OUTCOMES:
Gastrointestinal Symptoms in the Timecourse | Data are continuously collected from admission to discharge. Extraction occurs on the first three days of admission, weekly during the stay (on Mondays or Tuesdays, covering the preceding week), and on the final three days of discharge.
  The Gastrointestinal Symptom Rating Scale is assessed weekly during inpatient treament.
Dietary intake | Data are continuously collected throughout the inpatient stay. Extraction takes place on the day of admission, weekly during the stay (on Mondays or Tuesdays, reflecting the data of the preceding week), and on the day of discharge.
  Dietary intake is closely monitored from the beginning to the end of the inpatients stay. The data of the plans will be summarized weekly, containing information on the intake of macro- and micronutrients, fibre, energy intake and food groups. The outcome is analyzed seperately for patients with anorexia nervosa and bulimia nervosa.
Body weight | Data are continuously collected from admission to discharge. Extraction occurs the second day in the morning after admission, weekly during the stay (on Mondays or Tuesdays), and at the day of discharge
  Body weight in kg is measured in underwear in the morning before breakfast using a calibrated scale in order to calculate the Body mass index or body mass index z-score. The outcome is analyzed seperately for patients with anorexia nervosa and bulimia nervosa.
Body height | Body weight is measured within the first two days after admission and again within the final two days prior to discharge. For inpatient stays exceeding three months, weight measurements are repeated at three-month intervals.
  Body height in cm is measured using a standardized stadiometer to calculate the body mass index or the body mass index z-score. The outcome is analyzed seperately for patients with anorexia nervosa and bulimia nervosa.
Body composition | Body composition is measured within the first two days after admission and again within the final two days prior to discharge. The outcome is analyzed seperately for patients with anorexia nervosa and bulimia nervosa.
  Body composition is measured with bioelectrical impedance
Eating Disorder Inventory-2 (EDI-2) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  Eating Disorder Inventory-2 (EDI-2): A 91-item self-report questionnaire assessing psychological and behavioral traits related to eating disorders across 11 subscales. Each item is scored from 0 to 2; total scores range from 0 to 182, with higher scores indicating worse outcomes (greater symptom severity. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Three Factor Eating Questionnaire (TFEQ) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is a self-report measure of eating behavior with 51 items across three subscales: Cognitive Restraint, Disinhibition, and Hunger. Items are primarily dichotomous (yes/no), with some Likert-scale items. Subscale scores vary in range, and the total score ranges from 0 to 51, with higher scores indicating worse outcomes (e.g., more disinhibited eating, greater hunger, or excessive restraint). Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Symptom-Checkliste (SCL-90-R) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  Symptom-Checklist-90-Revised (SCL-90-R): A 90-item self-report questionnaire assessing general psychological distress across 9 symptom dimensions (e.g., depression, anxiety, somatization) and 3 global indices. Each item is rated from 0 (not at all) to 4 (extremely). Total scores range from 0 to 360, with higher scores indicating worse psychological symptom severity. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Beck-Depressions-Inventar Revision (BDI-II) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is a 21-item self-report questionnaire assessing the severity of depressive symptoms over the past two weeks. Each item is rated on a scale from 0 to 3. Total scores range from 0 to 63, with higher scores indicating worse depressive symptom severity. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Obsessive Compulsive Inventory - Revised (OCI-R) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is an 18-item self-report questionnaire measuring the severity of obsessive-compulsive symptoms across 6 subscales (e.g., washing, checking, hoarding). Each item is rated from 0 (not at all) to 4 (extremely). Total scores range from 0 to 72, with higher scores indicating worse obsessive-compulsive symptom severity. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Generalizied Anxiety Disorder Scale-7 (GAD-7) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is a 7-item self-report questionnaire assessing symptoms of generalized anxiety over the past two weeks. Each item is rated from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21, with higher scores indicating worse anxiety symptom severity. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Wender Utah Rating Scale (WURS-K) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is a 25-item self-report questionnaire assessing retrospective childhood symptoms of ADHD in adults. Each item is rated from 0 (not at all or never) to 4 (very much or very often). Total scores range from 0 to 100, with higher scores indicating greater severity of ADHD-related childhood symptoms. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Subthreshold Autism Trait Questionnaire (SATQ) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is a 24-item self-report questionnaire measuring the presence of subclinical autistic traits in adults. Each item is rated from 0 (strongly disagree) to 3 (strongly agree). Total scores range from 0 to 72, with higher scores indicating more pronounced subthreshold autistic traits.Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Frost Multidi-mensional Perfectionism Scale (FMPS) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is a 35-item self-report questionnaire assessing perfectionism across multiple dimensions, including concern over mistakes, personal standards, and parental expectations. Each item is rated from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 35 to 175, with higher scores indicating greater levels of perfectionism. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Perceived Stress Questionnaire (PSQ) | Data are collected within the first three days after admission and during the final three days before discharge (two time points).
  This is a self-report instrument assessing subjective experiences of stress over the past weeks. The standard version includes 30 items, each rated on a scale from 1 (almost never) to 4 (usually). Total scores range from 30 to 120, with higher scores indicating greater perceived stress. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Age | This is assessed upon admission.
  Age is assessed by documenting the birth date (day, months, year) from the health insurance card.
Complete Blood Count (CBC) with Differential | Data will be analyzed from samples collected within the first 3 days after hospital admission, weekly throughout the inpatient stay (on or around Day 7, Day 14, etc.), and within the final 3 days prior to discharge.
  Complete Blood Count (CBC) with Differential: A standard laboratory test used to assess general health and detect hematological abnormalities. Measures include red blood cells, white blood cells, hemoglobin, hematocrit, platelets, and a differential count of white blood cell subtypes (neutrophils, lymphocytes, monocytes, eosinophils, basophils). Results outside reference ranges may indicate infection, anemia, inflammation, or immune response abnormalities. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Key electrolyte panel for fluid balance, neuromuscular function, and metabolic regulation | Data will be analyzed from samples collected within the first 3 days after hospital admission, weekly throughout the inpatient stay (on or around Day 7, Day 14, etc.), and within the final 3 days prior to discharge.
  A standard blood chemistry panel measuring key electrolytes involved in fluid balance, neuromuscular function, and metabolic regulation.
  Sodium (Na⁺): typically 135-145 mmol/L
  Potassium (K⁺): typically 3.5-5.0 mmol/L
  Chloride (Cl-): typically 98-107 mmol/L
  Magnesium (Mg²⁺): typically 0.7-1.0 mmol/L
  Phosphate (PO₄³-): typically 0.8-1.5 mmol/L Abnormal values may indicate renal dysfunction, metabolic imbalance, or effects of medications. Higher or lower levels indicate worse physiological regulation depending on the parameter. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Liver Function Panel | Data will be analyzed from samples collected within the first 3 days after hospital admission, weekly throughout the inpatient stay (on or around Day 7, Day 14, etc.), and within the final 3 days prior to discharge.
  This Liver Function Panel (ALT, AST, GGT, ALP, Bilirubin, Albumin, INR) is a comprehensive blood test panel assessing hepatocellular injury and liver synthetic function.
  Alanine aminotransferase (ALT): < 50 U/L
  Aspartate aminotransferase (AST): < 50 U/L
  Gamma-glutamyl transferase (GGT): < 60 U/L
  Alkaline phosphatase (ALP): 35-125 U/L
  Total Bilirubin: 0.3-1.2 mg/dL
  Albumin: 3.5-5.0 g/dL
  International Normalized Ratio (INR): 0.9-1.2 Elevated enzyme levels may indicate hepatocellular injury or cholestasis, while changes in bilirubin, albumin, or INR reflect impaired liver function. Deviations from normal values indicate worsening liver status, depending on the parameter. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Renal Function Panel | Data will be analyzed from samples collected within the first 3 days after hospital admission, weekly throughout the inpatient stay (on or around Day 7, Day 14, etc.), and within the final 3 days prior to discharge.
  This Renal Function Panel (Creatinine, Urea/BUN, eGFR) is a standard blood test panel assessing kidney function and glomerular filtration.
  Serum Creatinine: typically 0.6-1.3 mg/dL
  Blood Urea Nitrogen (BUN)/Urea: typically 7-20 mg/dL (or 2.5-7.1 mmol/L)
  Estimated Glomerular Filtration Rate (eGFR): > 90 mL/min/1.73 m² (normal) Abnormal values may indicate impaired renal function, dehydration, or nephrotoxic effects. Higher creatinine or BUN and lower eGFR indicate worse kidney function. Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.
Medication Use | Data will be analyzed from samples collected within the first 3 days after hospital admission, weekly throughout the inpatient stay (on or around Day 7, Day 14, etc.), and within the final 3 days prior to discharge.
  Self-reported and/or medically verified use of prescribed or over-the-counter medications during the study period, with a focus on agents affecting gastrointestinal physiology. Values are recorded categorically (e.g., no medication, antidepressants, antipsychotics, anxiolytics, GI-active drugs, other). Data are analyzed separately for patients with anorexia nervosa and bulimia nervosa.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mack, Prof., Principal Investigator — University Hospital Tuebingen, Internal Medicine VI, Dept. of Psychosomatic Medicine and Psychotherapy
Locations (1):
- Klinik Lüneburger Heide, Bad Bevensen, Germany

IPD SHARING:
Plan to Share IPD: No
Patient data. Potential collaborators should contact us directly.

REFERENCES:
- [Background] Ketel J, Bosch-Bruguera M, Auchter G, Cuntz U, Zipfel S, Enck P, Mack I. Gastrointestinal Microbiota & Symptoms of Depression and Anxiety in Anorexia Nervosa-A Re-Analysis of the MICROBIAN Longitudinal Study. Nutrients. 2024 Mar 19;16(6):891. doi: 10.3390/nu16060891. PMID 38542802
- [Background] Mack I, Cuntz U, Gramer C, Niedermaier S, Pohl C, Schwiertz A, Zimmermann K, Zipfel S, Enck P, Penders J. Weight gain in anorexia nervosa does not ameliorate the faecal microbiota, branched chain fatty acid profiles, and gastrointestinal complaints. Sci Rep. 2016 May 27;6:26752. doi: 10.1038/srep26752. PMID 27229737
- [Background] Riedlinger C, Schmidt G, Weiland A, Stengel A, Giel KE, Zipfel S, Enck P, Mack I. Which Symptoms, Complaints and Complications of the Gastrointestinal Tract Occur in Patients With Eating Disorders? A Systematic Review and Quantitative Analysis. Front Psychiatry. 2020 Apr 20;11:195. doi: 10.3389/fpsyt.2020.00195. eCollection 2020. PMID 32425816
- [Background] Riedlinger C, Mazurak N, Schaffeler N, Stengel A, Giel KE, Zipfel S, Enck P, Mack I. Gastrointestinal complaints in patients with anorexia nervosa in the timecourse of inpatient treatment. Front Psychiatry. 2022 Aug 18;13:962837. doi: 10.3389/fpsyt.2022.962837. eCollection 2022. PMID 36061281